CLINICAL TRIAL: NCT04471337
Title: An Open-label Study to Evaluate the Pharmacokinetics and Safety of BAY 1817080 in Participants With Impaired Renal Function in Comparison to Matched Controls With Normal Renal Function
Brief Title: Study on the Safety of BAY1817080 How it is Tolerated and the Way the Body Absorbs, Distributes and Gets Rid of the Study Drug Given to Participants With Moderate Renal Impairment and End Stage Renal Disease Requiring Dialysis Compared With Matched Participants With Normal Renal Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 20332
Record Dates: First submitted 2020-07-10; First posted 2020-07-15 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Endometriosis Related Pain; Overactive Bladder; Diabetic Neuropathic Pain; Refractory or Unexplained Chronic Cough
Keywords: Normal renal function; Moderate renal impairment; End stage renal disease (ESRD); Dialysis
MeSH Terms: conditions — Urinary Bladder, Overactive; Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Arm A: Moderately impaired renal function (Experimental): Participants with moderately impaired renal function will receive multiple doses of BAY1817080.
  Interventions: Drug: BAY1817080
- Arm B: Normal renal function matched to Arm A (Experimental): Participants with normal renal function matched to Arm A will receive multiple doses of BAY1817080.
  Interventions: Drug: BAY1817080
- Arm C: End stage renal disease on dialysis (Experimental): Participants with ESRD requiring dialysis will receive single dose of BAY1817080.
  Interventions: Drug: BAY1817080
- Arm D: Normal renal function matched to Arm C (Experimental): Participants with normal renal function matched to Arm C will receive single dose of BAY1817080.
  Interventions: Drug: BAY1817080

INTERVENTIONS:
Drug: BAY1817080 — BAY1817080 will be administered orally as tablet.

SUMMARY:
BAY1817080 is currently under clinical development to treat pain related to unexplained chronic cough or chronic cough not affected by a treatment (refractory and/or unexplained chronic cough, RUCC), or a condition where the bladder is unable to hold urine normally (overactive bladder, OAB) or a condition in which tissue similar to the tissue that normally lines the inside of the womb grows outside the womb (endometriosis). Especially in elderly patients with OAB or RUCC, renal impairment is frequent. Renal impairment which co-occurs in especially in elderly patients with OAB or RUCC is a common condition in which the kidneys are not filtering the blood as well as they should. End stage renal disease (ESRD) requiring hemodialysis is a condition in which patients kidneys are no longer able to work as they should and require treatment to filter wastes from the blood. The goal of the study is to learn more about the safety of BAY1817080, how it is tolerated and the way the body absorbs, distributes and excretes the study drug given in men and women with moderate renal impairment and with those who have end stage renal disease (ESRD) requiring dialysis compared with matched participants with normal kidney function.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be 18 to 79 years of age inclusive, at the time of signing the informed consent.
* For renally impaired participants:

  * Decreased renal function, as assessed based on serum creatinine collected 2 to 10 days prior to dosing and calculated according to the Chronic Kidney Disease Epidemiology Collaboration formula (CKD-EPI) either: Moderately impaired renal function: eGFR: 30 to 59 mL/min/1.73 m^2; or ESRD on dialysis.
  * Stable renal disease, i.e. a serum creatinine value determined 3 or more months before screening (e.g. during routine diagnostics) should not differ by more than 25% from the serum creatinine value determined at screening.
* For participants with normal renal function:

  -- Normal renal function, as assessed at screening and based on serum creatinine according to the CKD-EPI : eGFR ≥90 mL/min/1.73 m^2.
* Body mass index (BMI) within the range 18 to 38 kg/m^2 (both inclusive)
* Women of childbearing potential (WOCBP) must agree to use contraception for the duration of the study. This applies for the time period between signing of the Informed Consent Form until at least 30 days after the last dose of the study drug.
* Capable of giving signed informed consent as described in study protocol which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.

Exclusion Criteria:

* Any relevant disease (other than those related to renal impairment for the renal impaired participants) within 4 weeks prior to study drug administration including infections and acute gastro-intestinal diseases (vomiting, diarrhea, constipation) requiring medical treatment.
* Acute renal failure or acute nephritis within the past 2 years
* Use of strong CYP3A4 and P-glycoprotein inhibitors from 2 weeks before study treatment until last day of blood sampling for pharmacokinetics after study drug administration.
* Use of CYP3A4 and P-glycoprotein inducers from 2 weeks before study treatment until last day of blood sampling for pharmacokinetics after study drug administration.
* Use of drugs which may affect absorption (e.g. loperamide, metoclopramide), and systemic administration of any broad-spectrum antibiotic within 1 week before first study drug administration, unless the drug is part of the mandatory dosing regimen for treatment of renal impairment or related conditions.
* International Normalized Ratio (INR) > 2.3.
* Indication or evidence for long QT syndrome; Participants in control group only: QT interval corrected using Fridericia's method (QTcF) > 450 msec.
* Inability to provide informed consent: Participants with psychiatric disorders.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2020-08-12 (Actual); Primary Completion 2021-02-15 (Actual); Study Completion 2021-05-06 (Actual)

PRIMARY OUTCOMES:
AUCu after single dose of BAY1817080 | On Day 1
  AUCu: Area under the Curve unbound
Cmax,u after single dose of BAY1817080 | On Day 1
  Cmax,u: maximum observed drug concentration in measured matrix after single dose administration (unbound)

SECONDARY OUTCOMES:
Number of subjects with treatment emergent adverse events (TEAEs) | From dosing up to 14 days after end of treatment with study medication
AUC (0-12)md,u after multiple dose of BAY1817080 | From Day 6 to Day 13
  Area under the time curve from 0-12 hours at steady state for the multiple dose (unbound)
Cmax,md,u after multiple dose of BAY1817080 | From Day 6 to Day 13
  Cmax,md,u: Maximum observed drug concentration at steady state for multiple dose (unbound)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Clinical Pharmacology of Miami, LLC, Miami, Florida
  - Orlando Clinical Research Center, Orlando, Florida

IPD SHARING:
Plan to Share IPD: No
There are no current plans to share data. Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.

REFERENCES:
- See also: Click here to find information for studies related to Bayer products. To find this study enter the ClinicalTrials.gov identifier (NCT) number or Bayer Study Identifier (ID) in the search field. — http://clinicaltrials.bayer.com/